CLINICAL TRIAL: NCT01896297
Title: A Prospective, Open Label Study to Evaluate the Pharmacokinetics of Dabigatran in Non-valvular Atrial Fibrillation (NVAF) Patients With Severely Impaired Renal Function on Dabigatran Etexilate 75 mg BID Therapy
Brief Title: Pradaxa Study in Non-valvular Atrial Fibrillation Patients With Severely Impaired Renal Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1160.173
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Results first posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran

ARMS (1):
- dabigatran etexilate (Other): 75mg BID by oral
  Interventions: Drug: Pradaxa, dabigatran etexilate

INTERVENTIONS:
Drug: Pradaxa, dabigatran etexilate — 75mg BID by oral

SUMMARY:
The goal of this study is to assess dabigatran pharmacokinetics in NVAF subjects with severe renal impairment defined as creatinine clearance between 15 and 30 mL/min calculated by Cockcroft-Gault formula.

The dabigatran etexilate dose of 75 mg BID was approved by the FDA for NVAF patients with severe renal impairment (CrCl 15-30 mL/min) , based on pharmacokinetic modeling and simulation.

ELIGIBILITY:
Inclusion criteria:

* Subjects diagnosed with non-valvular atrial fibrillation with an indication for the anticoagulation therapy,
* Subjects with severe renal function impairment defined as creatinine clearance between 15 and 30 mL/min by Cockcroft-Gault formula,
* Male and female patients, age =18 years at entry

Exclusion criteria:

* Contraindications to Pradaxa (history of a serious hypersensitivity reaction to Pradaxa, active pathological bleeding, patients with mechanical prosthetic heart valve),
* Creatinine clearance <15ml/min or patients with End Stage Renal Disease on dialysis,
* Creatinine clearance >30 ml/min,
* Pre-menopausal women (last menstruation less than one year prior to informed consent) who are nursing or pregnant, or are of child bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study. Acceptable methods of birth control include abstinence, tubal ligation, transdermal patch, intra uterine devices/systems (IUDs/IUSs), oral, implantable or injectable contraceptives, double barrier method and vasectomised partner,
* Patients who are participating in another drug study,
* Patients who have participated in another drug study within 6 weeks,
* Patients considered unreliable by the investigator concerning the requirements for participating in the study, including a follow-up interview,
* Any condition the investigator believes would not allow safe participation in the study,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (26):
- United States (26):
  - 1160.173.002 Boehringer Ingelheim Investigational Site, Hot Springs, Arkansas
  - 1160.173.023 Boehringer Ingelheim Investigational Site, Fremont, California
  - 1160.173.032 Boehringer Ingelheim Investigational Site, Moreno Valley, California
  - 1160.173.034 Boehringer Ingelheim Investigational Site, Oceanside, California
  - 1160.173.025 Boehringer Ingelheim Investigational Site, Salinas, California
  - 1160.173.033 Boehringer Ingelheim Investigational Site, San Pedro, California
  - 1160.173.024 Boehringer Ingelheim Investigational Site, Wilmington, Delaware
  - 1160.173.010 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 1160.173.020 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1160.173.036 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1160.173.012 Boehringer Ingelheim Investigational Site, Largo, Florida
  - 1160.173.013 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1160.173.005 Boehringer Ingelheim Investigational Site, Columbus, Georgia
  - 1160.173.018 Boehringer Ingelheim Investigational Site, Springfield, Missouri
  - 1160.173.019 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1160.173.026 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1160.173.027 Boehringer Ingelheim Investigational Site, Neptune City, New Jersey
  - 1160.173.014 Boehringer Ingelheim Investigational Site, Wilmington, North Carolina
  - 1160.173.001 Boehringer Ingelheim Investigational Site, Altoona, Pennsylvania
  - 1160.173.008 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1160.173.037 Boehringer Ingelheim Investigational Site, Lancaster, South Carolina
  - 1160.173.030 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 1160.173.011 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 1160.173.006 Boehringer Ingelheim Investigational Site, Live Oak, Texas
  - 1160.173.021 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 1160.173.035 Boehringer Ingelheim Investigational Site, Waukesha, Wisconsin

REFERENCES:
- [Derived] Martin JL, Esmaeili H, Manuel RC, Petrini M, Wiebe S, Maas H. Pharmacokinetics/Pharmacodynamics of Dabigatran 75 mg Twice Daily in Patients With Nonvalvular Atrial Fibrillation and Severely Impaired Renal Function. J Cardiovasc Pharmacol Ther. 2018 Sep;23(5):399-406. doi: 10.1177/1074248418769167. Epub 2018 Apr 25. PMID 29695165

RESULTS

PARTICIPANT FLOW:
Groups:
- Dabigatran Etexilate: Dabigatran etexilate 75mg capsule administered orally, twice daily (BID), for at least 7 days.
Period: Overall Study
Arm/Group | Dabigatran Etexilate
Started | 60
Completed | 59
Not Completed | 1
Not completed — Died in post treatment phase | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS) which included all enrolled patients who were eligible to enter the trial, who were dispensed trial medication and were documented to have taken at least one dose of trial drug.
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 83.35 (7.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Pre-dose Concentration of the Analyte in Plasma at Steady State Immediately Before Administration of the Next Dose
Description: Pre-dose concentration of the analyte in plasma at steady state immediately before administration of the next dose (Cpre,ss) taken at approximately 12 hours after the last dose (trough).
Time Frame: Immediately before the last drug administration, on day 8
Population: Pharmacokinetic (PK) set (PKS) which included all patients in the treated set with analyzable data in at least one observation for at least one primary endpoint without important protocol violations relevant to the evaluation of PK. Analysis includes patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 51
ng/mL | 155 (76.9)

2. Primary Outcome: Concentration of Analyte in Plasma at Steady State at 2 Hours After Administration of the Last Dose
Description: Concentration of analyte in plasma at steady state at 2 hours after administration of the last dose (C2,ss)
Time Frame: 2 hours after the last drug administration, on day 8
Population: PKS. Analysis includes patients with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 59
ng/mL | 202 (70.6)

ADVERSE EVENTS:
Time Frame: From first drug administration until 3 days after last drug administration, up to 18 days
Arm/Group | Dabigatran Etexilate
Serious Adverse Events (participants affected / at risk) | 2/60
Other Adverse Events (participants affected / at risk) | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate (N=60)
Acute myocardial infarction (Cardiac disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.